CLINICAL TRIAL: NCT03789877
Title: Enhancing A Home-Based Walking Intervention Among Breast Cancer Survivors With rTMS: Feasibility and Limited Efficacy Testing
Brief Title: A Home-Based Walking Program and rTMS in Helping Breast Cancer Survivors Get More Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: I 72218; NCI-2018-03302 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 72218 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-12-26; First posted 2018-12-31 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Cancer Survivor; Invasive Breast Carcinoma
MeSH Terms: interventions — Exercise; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (home-based walking program, rTMS) (Experimental): Patients participate in a home-based exercise program of at least 10,000 steps per day (about 30 minutes of daily exercise) for 5 days weekly (150 minutes per week) for 12 weeks. Patients also undergo repetitive transcranial magnetic stimulation over 1 hour for 8 sessions during the first 2 weeks of the walking program.
  Interventions: Other: Physical Activity; Other: Questionnaire Administration; Procedure: Repetitive Transcranial Magnetic Stimulation
- Group II (home-based exercise program, sham rTMS) (Active Comparator): Patients participate in a home-based exercise program of at least 10,000 steps per day (about 30 minutes of daily exercise) for 5 days weekly (150 minutes per week) for 12 weeks. Patients also undergo sham repetitive transcranial magnetic stimulation over 1 hour for 8 sessions during the first 2 weeks of the walking program.
  Interventions: Other: Physical Activity; Other: Questionnaire Administration; Procedure: Sham Intervention

INTERVENTIONS:
Other: Physical Activity — Participate in home-based walking program
Other: Questionnaire Administration — Ancillary studies
Procedure: Repetitive Transcranial Magnetic Stimulation — Undergo rTMS
  Other Names: rTMS
  Arms: Group I (home-based walking program, rTMS)
Procedure: Sham Intervention — Undergo sham rTMS
  Arms: Group II (home-based exercise program, sham rTMS)

SUMMARY:
This trial studies how well a home-based walking program, with or without repetitive transcranial magnetic stimulation, works in helping breast cancer survivors get more physical activity. Physical activity has been shown to improve health outcomes and quality of life among breast cancer survivors and can help lessen certain side effects of treatment such as fatigue, depression, and treatment-related weight gain. Repetitive transcranial magnetic stimulation is a procedure that uses electromagnets to stimulate brain activity. Using rTMS with a home-based walking program may help breast cancer survivors get more physical activity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the effects of 20 hertz (Hz) repetitive transcranial magnetic stimulation (rTMS) on delay discounting rates and multiple measures of self-regulation and walking.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients participate in a home-based exercise program of at least 10,000 steps per day (about 30 minutes of daily exercise) for 5 days weekly (150 minutes per week) for 12 weeks. Patients also undergo repetitive transcranial magnetic stimulation over 1 hour for 8 sessions during the first 2 weeks of the walking program.

GROUP II: Patients participate in a home-based exercise program of at least 10,000 steps per day (about 30 minutes of daily exercise) for 5 days weekly (150 minutes per week) for 12 weeks. Patients also undergo sham repetitive transcranial magnetic stimulation over 1 hour for 8 sessions during the first 2 weeks of the walking program.

ELIGIBILITY:
Inclusion Criteria:

* Have a previous history of invasive breast cancer who have completed treatment, except for hormonal therapy.
* Approved by a participant's physician to participate in this study.
* Have a smart phone or tablet with the capability of downloading the Fitbit activity tracker application, and a willingness to sync Fitbit activity tracker data with the application daily.
* Right handed.
* Pass the Transcranial Magnetic Stimulation Adult Safety and Screening questionnaire (TASS).
* Ability to speak and read English.

Exclusion Criteria:

* Pregnant or nursing.
* Have metastatic breast cancer.
* Morbidly obese as defined by a body mass index (BMI) >= 40.
* Have any condition which would preclude receiving rTMS, including:

  * Personal history of epilepsy, head injury, aneurysm, stroke, or previous cranial neurosurgery or abnormal findings on the MRI (e.g., tumor, aneurysm, etc.)
  * A self-reported diagnosis of major depressive disorder, bipolar disorder or a schizophrenia-spectrum disorder, or tinnitus.
  * Metal implants or neuro-stimulators in the head, neck, or cochlea.
  * A pacemaker.
  * Known pre-existing noise induced hearing loss or concurrent treatment with ototoxic medications (i.e., aminoglycosides, cisplatin).
  * Use of anticonvulsant medication, or currently taking medications that lower seizure threshold (e.g., such as tricyclic antidepressants or bupropion).
  * Participants who score above 48.3 on the Claustrophobia questionnaire at the baseline assessment will be excluded because they are likely to be unable to undergo an Magnetic Resonance Imaging (MRI) without distress.
* Unwilling or unable to follow protocol requirements.
* Any condition which the principal investigator determines will make the participant an unsuitable candidate to participate in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Delay discounting score | Baseline up to 6 months
  The effect of the transcranial magnetic stimulation (TMS) intervention on the delay discounting score will be assessed using a two-arm, randomized, double-blind, sham controlled repeated measures design. The efficacy of TMS will be quantified by comparing the within-patient change in delay discounts scores between the baseline and week 12 assessments in the evaluable sample. The treatment effect will be estimated with a generalized linear mixed model, describing the continuous delay discounting outcomes as a function of a random participant effect, and fixed effects for treatment assignment (TMS reference: sham), categorical visit number (4 levels), and the treatment/visit interaction. The magnitude, direction and 95% confidence interval for the adjusted interaction term estimate will be used to describe the effect of TMS on the delay discounting score. These results will be supported by descriptive statistics and graphical depictions of the results as appropriate.
Number of steps per day | Baseline up to 6 months
  The effects of TMS on steps per day will be quantified by comparing the within-patient change in these outcomes between the baseline and week 12 assessments in the evaluable sample. The treatment effect will be estimated with a generalized linear mixed model as described above. These results will be supported by descriptive statistics and graphical depictions of the results as appropriate. This analysis will be used to determine the feasibility of using rTMS to enhance a home-based walking intervention among breast cancer survivors, based on whether breast cancer survivors who receive active rTMS demonstrate more steps per day than breast cancer survivors who receive sham rTMS.
Number of minutes of moderate physical activity per day | Baseline up to 6 months
  The effects of TMS on minutes of activity per week will be quantified by comparing the within-patient change in these outcomes between the baseline and week 12 assessments in the evaluable sample. The treatment effect will be estimated with a generalized linear mixed model as described above. These results will be supported by descriptive statistics and graphical depictions of the results as appropriate. This analysis will be used to determine the feasibility of using rTMS to enhance a home-based walking intervention among breast cancer survivors, based on whether breast cancer survivors who receive active rTMS demonstrate more minutes of moderate intensity activity than breast cancer survivors who receive sham rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sheffer, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States